CLINICAL TRIAL: NCT05946512
Title: MR Spectroscopy in Well-characterized Individuals With and Without Post COVID Condition Prior to and Following a Yoga Breathing Intervention- an Explorative Randomised Controlled Trial
Brief Title: MR-spectroscopy in Post-covid Condition Prior to and Following a Yoga Breathing Intervention
Acronym: SpeCY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1034/2023
Record Dates: First submitted 2023-07-13; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Post COVID-19 Condition; Somatic Symptom Disorder
Keywords: Yoga breathing intervention; dysfunctional breathing; MR-Spectroscopy
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga intervention (Experimental)
  Interventions: Behavioral: yoga
- social contact (Active Comparator)
  Interventions: Behavioral: social contact

INTERVENTIONS:
Behavioral: yoga — yoga breathing techniques for dysfunctional breathing
  Arms: yoga intervention
Behavioral: social contact — social contact as active comparator
  Arms: social contact

SUMMARY:
From a clinical perspective, we find that many patients with Post COVID condition suffer from severe and debilitating shortness of breath, while routine pulmonary investigations fail to find the cause of the problems experienced. If dyspnea is associated with palpitations, dizziness or anxiety, patients are commonly diagnosed with "dysfunctional breathing". From a psychosomatic perspective, the symptom of dysfunctional breathing can be classified as a "functional symptom" under the umbrella term of somatic symptom disorder. Therefore, Yoga interventions with special emphasis on breath-guided relaxation are a promising approach. We aim to investigate the psycho-somatic and somato-psychic pathophysiology on a morphological, psychological, functional and biological basis underlying the symptom of dysfunctional breathing. Furthermore, we plan to investigate the mechanism of Yoga intervention on the mental and somatic symptom burden of participants with Post COVID condition. Then, we aim to compare the impact of Yoga on other groups - healthy individuals, patients with chronic obstructive lung disease (COPD), as well as those with somatic symptom disorder. As a control intervention to Yoga guided breathing exercises a social contact group will be used.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for participants with Post COVID condition

  1. Eligible patients will be recruited at the Respiratory Outpatient Clinic (Medical University Innsbruck, Internal Medicine II) from the PRECISE registry or from other participating clinics at Medical University Innsbruck and via local advertisement.
  2. Persistent respiratory symptoms for 3 months after infection (mMRC dyspnea score ≥ 1).
  3. Absence of obstructive or restrictive lung disease or unilateral diaphragmatic paresis.
  4. Medical history with symptoms compatible with DB as assessed by the physician AND Nijmegen cut-off score of >23 or reduced MIP. The last two conditions were chosen to provide a readily accessible and objectifiable entry criterion at the inclusion visit.
  5. Age >= 18 years, < 50 years.
  6. Sufficient knowledge of German language for interaction during Yoga and completion of questionnaires.

Inclusion criteria for participants with COPD

1. Eligible patients will be recruited at the Respiratory Outpatient Clinic (Medical University Innsbruck).
2. A postbronchodilator FEV1/FVC ratio less than 0,7 obtained in functional pulmonary testing is required fo diagnosis of COPD (Global Initiative for Chronic Obstructive Lung Disease (GOLD) Science Committee, 2022).
3. Persistent respiratory symptoms for 3 months (mMRC≥ 1).
4. Absence of unilateral diaphragmatic paresis.
5. Medical history with symptoms compatible with DB as assessed by the physician AND Nijmegen cut-off score of >23 or reduced MIP. The last two conditions were chosen to provide a readily accessible and objectifiable entry criterion at the inclusion visit.
6. Age >= 18 years, < 50 years
7. Sufficient knowledge of German language for interaction during Yoga and completion of questionnaires

Inclusion criteria for participants with somatic symptom disorder

1. Eligible patients will be recruited at University Hospital for Psychiatry I and II, Medical University Innsbruck) and via local advertisement.
2. Screening positive for somatic symptoms disorder with the following scores: SSD-12 ≥ 23, SSS-8 ≥ 9.
3. Persistent respiratory symptoms for 3 months after infection (mMRC≥ 1).
4. Absence of obstructive or restrictive lung disease or unilateral diaphragmatic paresis.
5. Absence of medical history with symptoms compatible with DB as assessed by the physician AND Nijmegen cut-off score of >23 or reduced MIP. The last two conditions were chosen to provide a readily accessible and objectifiable entry criterion at the inclusion visit.
6. Age >= 18 years, < 50 years.
7. Sufficient knowledge of German language for interaction during Yoga and completion of questionnaires.

Inclusion criteria for healthy participants

1. Eligible participants will be recruited via local advertisement.
2. Absence of significant active mental or somatic disorders
3. Absence of persistent respiratory symptoms (mMRC< 1).
4. Absence of obstructive or restrictive lung disease or unilateral diaphragmatic paresis.
5. Absence of medical history with symptoms compatible with DB as assessed by the physician AND Nijmegen questionnaire and MIP within normal limits..
6. Age >= 18 years, < 50 years.
7. Sufficient knowledge of German language for interaction during Yoga and completion of questionnaires.

Exclusion Criteria:

* Exclusion criteria for participants with post COVID condition

  1. Conditions precluding magnetic resonance imaging (MRI) such as metal implants in the body (e.g., pacemakers, surgical devices), phobic anxiety, claustrophobia, or pregnancy.
  2. Active psychiatric conditions interfering with study participation such as psychosis or acute suicidality.
  3. Severe fatigue interfering with study participation.
  4. Previous evidence of structural brain abnormality on the structural MRI scan.
  5. Significant previous meditation or Yoga experience.
  6. Patients with known carotid stenosis >70% or cardiopulmonary contraindications for tilt table and other cardiovascular autonomic function tests (e.g. Valsalva maneuver, deep breathing, standing test).

Exclusion criteria for participants with COPD

1. Conditions precluding magnetic resonance imaging (MRI) such as metal implants in the body (e.g., pacemakers, surgical devices), phobic anxiety, claustrophobia, or pregnancy.
2. Active psychiatric conditions interfering with study participation such as psychosis or acute suicidality.
3. Severe fatigue interfering with study participation.
4. Previous evidence of structural brain abnormality on the structural MRI scan.
5. Medical history of post COVID condition.
6. Significant previous meditation or Yoga experience.
7. Patients with known carotid stenosis >70% or cardiopulmonary contraindications for tilt table and other cardiovascular autonomic function tests (e.g. Valsalva maneuver, deep breathing, standing test).
8. Patients dependent on a long-term oxygen therapy (LTOT )

Exclusion criteria for participants with somatic symptom disorder

1. Conditions precluding magnetic resonance imaging (MRI) such as metal implants in the body (e.g., pacemakers, surgical devices), phobic anxiety, claustrophobia, or pregnancy.
2. Other active psychiatric conditions interfering with study participation such as psychosis or acute suicidality.
3. Severe fatigue interfering with study participation.
4. Previous evidence of structural brain abnormality on the structural MRI scan.
5. Medical history of post COVID condition.
6. Significant previous meditation or Yoga experience.
7. Patients with known carotid stenosis >70% or cardiopulmonary contraindications for tilt table and other cardiovascular autonomic function tests (e.g. Valsalva maneuver, deep breathing, standing test).

Exclusion criteria for healthy participants

1. Conditions precluding magnetic resonance imaging (MRI) such as metal implants in the body (e.g., pacemakers, surgical devices), phobic anxiety, claustrophobia, or pregnancy.
2. Active psychiatric conditions interfering with study participation such as psychosis or acute suicidality.
3. Previous evidence of structural brain abnormality on the structural MRI scan.
4. Medical history of post COVID condition.
5. Significant previous meditation or Yoga experience.
6. Patients with known carotid stenosis >70% or cardiopulmonary contraindications for tilt table and other cardiovascular autonomic function tests (e.g. Valsalva maneuver, deep breathing, standing test).

legend: PRECISE = a study conducted with participants with post-COVID-19 condition at the Medical University of Innsbruck; mMRC score = modified medical research council score; DB = dysfunctional breathing; MIP = maximal inspiratory pressure; COPD = chronic obstructive pulmonary disease; FEV1/FVC = forced expiratory volume in one second/ forced vital capacity; SSD-12 = Somatic Symptom Disorder - B Criteria Scale; SSS-8 = Somatic Symptom Scale - 8;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-07-24 (Estimated); Primary Completion 2026-07-24 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
brain imaging | 10 weeks
  31P MRI

SECONDARY OUTCOMES:
comparison with control groups | 10 weeks
  resting state functional MRI (rs-MRI),diaphragmatic function in spirometry and MRI, laboratory analyses, autonomic testing, questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Universität Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No